CLINICAL TRIAL: NCT03034395
Title: Pilot Study of 1cm Versus 2cm Margins for the Surgical Treatment of cT2N0M0 Melanoma
Brief Title: Study of 1cm Versus 2cm Margins for the Surgical Treatment of cT2N0M0 Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2016-JM-MEL-T2Margins
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; cT2N0M0
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide Local Excision 1cm (Other)
  Interventions: Procedure: Wide Local Excision
- Wide Local Excision 2cm (Other)
  Interventions: Procedure: Wide Local Excision

INTERVENTIONS:
Procedure: Wide Local Excision — Surgery

SUMMARY:
This is a randomized non-blinded pilot study for patients with melanoma staging cT2N0M0 who are candidates for surgical resection. The primary objective is to determine the feasibility of randomizing participants with cT2N0M0 malignant melanoma to surgical treatment with 1cm versus 2cm margins. Study will try to determine overall survival for cT2N0M0 malignant melanoma after surgical treatment with 1cm versus 2cm margins.

DETAILED DESCRIPTION:
After randomization, participants will undergo surgery with wide local excision with either 1cm or 2cm margins. The margin will be based upon the previous biopsy site or area of pigmentation. The skin and subcutaneous tissue (down to fascia) will be resected. Closure considerations may require removal of additional tissue for non-oncologic purposes. As per standard of care, sentinel lymph node biopsy will be performed using a dual tracer technique (technetium radiolabeled sulfur colloid and isosulfan blue) with or without lymphoscintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven T2 malignant melanoma.
* Eastern Cooperative Oncology Group (ECOG) score of 0-2.

Exclusion Criteria:

* Visible additional disease that suggests a greater than T2 malignant melanoma
* Unable to tolerate general anesthesia
* Evidence of distant metastatic disease
* Melanoma located on face or digits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who agree to blinded randomization to a surgical margin trial for the treatment of early stage melanoma. | 2 years
  Number of patients who agree to participate

SECONDARY OUTCOMES:
Recurrence (disease free survival) | Every 4 months post-surgery for 2 years and then every 4-6 months for an additional 3 years
  Subjects will be evaluated at 4 month intervals for 2 years and then at 4-6 month intervals for an additional 3 years to evaluate for evidence of disease recurrence.
Quality of life following surgery | One month post-surgery
  Measured by FACT-Melanoma Surgery Subscale

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mammen, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States